CLINICAL TRIAL: NCT02803398
Title: Modelling Interface Pressure Applied by Superimposed Compression Bandages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A01219-40
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Risk of Venous Thrombosis
Keywords: Compression bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient at risk of venous thrombosis (Experimental)
  Interventions: Other: Compression bandages application and interface pressure measurements

INTERVENTIONS:
Other: Compression bandages application and interface pressure measurements — Bandages, which are applied in a spiral pattern on the leg, are composed of Biflex 16 (Thuasne) and/or Rosidal K (Lohmann & Rauscher).

SUMMARY:
The aim of the study is to measure and model interface pressure applied on the lower leg of patients at risk of veinous thrombosis, by different bandage combinations, composed of Biflex 16 (Thuasne) and/or Rosidal K (Lohmann & Rauscher). The patient specific model should better predict the interface pressure distribution than Laplace's Law.

DETAILED DESCRIPTION:
The measurement of the patients' legs shapes will be performed thanks to an optical scanner. The patients' posterior part of the calf will be submitted to a localized compression test, in order to characterize the soft tissue mechanical properties of both legs.

Pressure measurements, applied by the different bandages, will be taken at the height of measurement points B1 and C on the lateral and medial sides of the leg in supine, sitting and standing positions, on both legs.

2 single bandages (Biflex 16 (Thuasne) and Rosidal K (Lohmann & Rauscher)) and their different combinations will be applied on the patient's legs.

The order of bandage application for each patient is randomized, but is the same for both legs. The order of the leg (right or left) on which the bandages are applied is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 80 years old
* at risk of venous thrombosis, who need to wear compression (socks, stockings or bandage)
* Hospitalized in the Service of Physical Medicine and Rehabilitation, in Saint-Etienne, France
* BMI between 20 and 35
* Able to stand for at least 10 minutes in a standing frame
* Signed informed consent to take part in the study
* Covered by a health insurance system
* Not taking part in another study which interfere with the results of the present study

Exclusion Criteria:

* Compression bandages contraindications
* Allergy to one of the different bandages components
* History of deep or superficial vein thrombosis
* Venous or arterial ulcer
* Cutaneous wound on the lower leg
* Cognitive, behavior or physical disorder preventing the communication and the active participation to a rehabilitation program, or a clinical study
* Patient under any legal protection (except curatorship)
* Not covered by a health insurance system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Consistency between interface pressure [mmHg] given by the patient-specific simulation and the experimental pressure measurements for different positions (supine, sitting, standing) and the different bandage combinations. | Through study completion (one year)

SECONDARY OUTCOMES:
Evaluation of the impact of soft tissue mechanical propreties on interface pressure | Through study completion (one year)
  Patient's leg soft tissue mechanical properties are characterized for both patient's legs before bandage application. The impact of this parameter on the measured interface pressure will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Giraux, MD, PhD, Principal Investigator — Service de Médecine Physique et de Réadaptation, CHU Saint-Etienne, France
Locations (1):
- Service de Médecine Physique et de Réadaptation, CHU Bellevue, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chassagne F, Helouin-Desenne C, Molimard J, Convert R, Badel P, Giraux P. Superimposition of elastic and nonelastic compression bandages. J Vasc Surg Venous Lymphat Disord. 2017 Nov;5(6):851-858. doi: 10.1016/j.jvsv.2017.07.006. PMID 29037358